CLINICAL TRIAL: NCT03579459
Title: A PHASE 3, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLINDED STUDY TO EVALUATE THE LOT CONSISTENCY, SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A CLOSTRIDIUM DIFFICILE VACCINE IN HEALTHY ADULTS 65 TO 85 YEARS OF AGE
Brief Title: Evaluation Of Clostridium Difficile Vaccine Lot Consistency In Healthy Adults 65 To 85 Years Of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B5091008
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Clostridium Difficile Associated Disease
Keywords: Clostridium Difficile; vaccine
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Clostridium difficile vaccine Lot 1 (Active Comparator)
  Interventions: Biological: Clostridium difficile vaccine
- Clostridium difficile vaccine Lot 2 (Active Comparator)
  Interventions: Biological: Clostridium difficile vaccine
- Clostridium difficile vaccine Lot 3 (Active Comparator)
  Interventions: Biological: Clostridium difficile vaccine
- Placebo (Placebo Comparator): Normal saline solution (0.9% sodium chloride)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Clostridium difficile vaccine — Toxoid based Clostridium difficile vaccine
  Arms: Clostridium difficile vaccine Lot 1; Clostridium difficile vaccine Lot 2; Clostridium difficile vaccine Lot 3
Biological: placebo — Normal saline solution
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
This study will investigate a Clostridium difficile vaccine in healthy adults 65 to 85 years of age, who will each receive 3 doses of vaccine. The study will assess the lot consistency, safety, and tolerability of the vaccine, and also look at the subjects' immune response to the vaccine.

DETAILED DESCRIPTION:
Serology for B5091008 was delayed due to discussions with the FDA on statistical analysis as well as delays attributed to the COVID pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document.
* Willing and able to comply with study procedures.
* Healthy adults 65 to 85 years of age.
* Male subjects or female subjects who are not of childbearing potential.
* Ability to be contacted by telephone during study participation.

Exclusion Criteria:

* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s)/vaccine(s) within 28 days prior to study entry through conclusion of the study.
* Previous administration of an investigational C difficile vaccine or C difficile monoclonal antibody therapy.
* Proven or suspected prior episode of C difficile infection.
* Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 8 weeks before receipt of investigational product.
* Serious chronic medical disorders, including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease.
* Any bleeding disorder or anticoagulant therapy that would contraindicate intramuscular injection.
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components.
* Subjects who may be unable to respond to vaccination due to:

  * Congenital or acquired immunodeficiency.
  * Receipt of systemic corticosteroids (greater than or equal to 20 mg/day of prednisone or equivalent) for greater than or equal to 14 days within 28 days of enrollment.
  * Receipt of chronic systemic treatment with other known immunosuppressant medications, or radiotherapy, within 6 months of enrollment.
  * Underlying bone marrow disorder treated within the past year, such as myelodysplasia, myeloma, or myeloproliferative disorder, treated within the past year, or any history of bone marrow transplant.
  * Malignancy that required treatment with chemotherapy (including the use of adjunctive and hormonal therapy), immunotherapy, radiation therapy, or antineoplastic target therapies within the past 24 months.
* Receipt of blood products or immunoglobulins within 6 months before enrollment through conclusion of the study.
* Residence in a nursing home or other long-term care facility, or requirement for semiskilled nursing care or assisted living. An ambulatory subject who lives in an autonomous manner in a retirement home or village is eligible for the trial.
* A known infection with human immunodeficiency virus (HIV).
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavioral or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results.
* Female subjects of childbearing potential; pregnant female subjects; breastfeeding female subjects; fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1317 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (24):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Advanced Clinical Research, Meridian, Idaho
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Amici Clinical Research, Raritan, New Jersey
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Medical Research South, LLC, Goose Creek, South Carolina
  - Benchmark Research, Austin, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc./ Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Incorporated/Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Christensen S, Bouguermouh S, Ilangovan K, Pride MW, Webber C, Lockhart SP, Shah R, Kitchin N, Lamberth E, Zhang H, Gao Q, Brock L, Anderson AS, Gruber WC. A phase 3 study evaluating the lot consistency, immunogenicity, safety, and tolerability of a Clostridioides difficile vaccine in healthy adults 65 to 85 years of age. Vaccine. 2023 Dec 7;41(50):7548-7559. doi: 10.1016/j.vaccine.2023.11.003. Epub 2023 Nov 17. PMID 37977942
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5091008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1358 participants signed the informed consent form (ICF). 41 participants were screen failures who did not meet eligibility criteria and were not enrolled. Out of 1317 randomized participants, only 1314 participants received at least one 1 dose of the investigational product.
Groups:
- Clostridium Difficile Vaccine: Lot 1: Participants were randomized to receive Clostridium difficile vaccine Lot 1 (200 microgram total toxoid per dose) intramuscularly at Months 0, 1 and 6.
- Clostridium Difficile Vaccine: Lot 2: Participants were randomized to receive Clostridium difficile vaccine Lot 2 (200 microgram total toxoid per dose) intramuscularly at Months 0, 1 and 6.
- Clostridium Difficile Vaccine: Lot 3: Participants were randomized to receive Clostridium difficile vaccine Lot 3 (200 microgram total toxoid per dose) intramuscularly at Months 0, 1 and 6.
- Placebo: Participants were randomized to receive placebo (0.9% sodium chloride injection, in a 0.5 mL dose) intramuscularly at Months 0, 1 and 6.
Period: Overall Study
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Started | 330 | 327 | 328 | 332
Dose 1 | 330 | 325 | 328 | 331
Dose 2 | 324 | 318 | 319 | 322
Dose 3 | 305 | 305 | 307 | 309
Completed | 301 | 304 | 305 | 308
Not Completed | 29 | 23 | 23 | 24
Not completed — Adverse Event | 7 | 6 | 2 | 6
Not completed — Death | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 6 | 2 | 4 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 3 | 5
Not completed — Withdrawal by Subject | 12 | 8 | 11 | 8
Not completed — Medication error without associated adverse event | 2 | 1 | 1 | 0
Not completed — Other | 0 | 1 | 1 | 0
Not completed — Randomized not vaccinated | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product.
Groups:
- Clostridium Difficile Vaccine: Lot 1: Participants received Clostridium difficile vaccine Lot 1 (200 microgram total toxoid per dose) intramuscularly at Months 0, 1 and 6.
- Clostridium Difficile Vaccine: Lot 2: Participants received Clostridium difficile vaccine Lot 2 (200 microgram total toxoid per dose) intramuscularly at Months 0, 1 and 6.
- Clostridium Difficile Vaccine: Lot 3: Participants received Clostridium difficile vaccine Lot 3 (200 microgram total toxoid per dose) intramuscularly at Months 0, 1 and 6.
- Placebo: Participants received placebo (0.9% sodium chloride injection, in a 0.5 mL dose) intramuscularly at Months 0, 1 and 6.
- Total: Total of all reporting groups
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo | Total
Number analyzed (Participants) | 330 | 325 | 328 | 331 | 1314
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (5.01) | 72.0 (5.03) | 71.1 (4.83) | 72.1 (4.99) | 71.7 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 186 | 186 | 178 | 739
  Male | 141 | 139 | 142 | 153 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 29 | 26 | 32 | 125
  Not Hispanic or Latino | 289 | 291 | 299 | 297 | 1176
  Unknown or Not Reported | 3 | 5 | 3 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 2 | 3 | 8
  Asian | 5 | 5 | 6 | 6 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 3 | 2 | 7
  Black or African American | 38 | 25 | 29 | 25 | 117
  White | 285 | 289 | 285 | 292 | 1151
  More than one race | 0 | 1 | 2 | 2 | 5
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Clostridium Difficile Toxin A and Toxin B Specific Neutralizing Antibodies at Month 7
Description: GMC was calculated as the mean of the assay results after making the logarithm transformation and then back transformation to its original scale. Confidence intervals (CIs) were back transformations of CIs based on the Student t distribution for the mean logarithm of the concentrations. Clostridium difficile toxin A and toxin B were inactivated by a combination of genetic mutations to decrease toxin activity and chemical treatments were done prior to final purification and formulation of the drug substance.
Time Frame: At Month 7
Population: Evaluable immunogenicity(EI)population=enrolled participants who received all 3 doses of investigational product to which they were randomized; blood drawn for analysis within 23-47 days after visit 4(Month 6)had valid, determinate assay results for either toxinA or B for specified analysis and no major protocol deviations. Placebo arm is not reported as GMC was planned to be evaluated only for 3 vaccine lots. Here,'Number Analyzed' refers to number of participants evaluable for specific toxins.
Measure: Geometric Mean (95% Confidence Interval); unit: Neutralization units per mL
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3
Number analyzed (Participants) | 286 | 284 | 296
Neutralization units per mL
  Toxin A: number analyzed (Participants) | 286 | 284 | 295
  Toxin A | 878.8 [786.3 to 982.2] | 873.0 [779.2 to 978.1] | 872.9 [782.6 to 973.5]
  Toxin B: number analyzed (Participants) | 285 | 283 | 296
  Toxin B | 5823.9 [5041.0 to 6728.4] | 5462.8 [4733.4 to 6304.7] | 5426.0 [4724.4 to 6231.8]
Statistical Analysis 1: Comparison: Clostridium Difficile Vaccine: Lot 1 vs Clostridium Difficile Vaccine: Lot 2; Toxin A; Test type: Equivalence — Equivalence was established if the 95% confidence interval of GMC ratio was within the interval (0.5, 2); Geometric Mean ratio (GMR) = 1.01, 95% CI 2-sided [0.86 to 1.18] — Confidence intervals (CIs) were back transformations of confidence levels based on the Student t distribution for the mean logarithm of the concentrations
Statistical Analysis 2: Comparison: Clostridium Difficile Vaccine: Lot 1 vs Clostridium Difficile Vaccine: Lot 3; Toxin A; Test type: Equivalence — Equivalence was established if the 95% confidence interval of GMC ratio was within the interval (0.5, 2); GMR = 1.01, 95% CI 2-sided [0.86 to 1.18] — CIs were back transformations of confidence levels based on the Student t distribution for the mean logarithm of the concentrations
Statistical Analysis 3: Comparison: Clostridium Difficile Vaccine: Lot 2 vs Clostridium Difficile Vaccine: Lot 3; Toxin A; Test type: Equivalence — Equivalence was established if the 95% confidence interval of GMC ratio was within the interval (0.5, 2); GMR = 1.00, 95% CI 2-sided [0.85 to 1.17] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Clostridium Difficile Vaccine: Lot 1 vs Clostridium Difficile Vaccine: Lot 2; Toxin B; Test type: Equivalence — Equivalence was established if the 95% confidence interval of GMC ratio was within the interval (0.5, 2); GMR = 1.07, 95% CI 2-sided [0.87 to 1.31] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Clostridium Difficile Vaccine: Lot 1 vs Clostridium Difficile Vaccine: Lot 3; Toxin B; Test type: Equivalence — Equivalence was established if the 95% confidence interval of GMC ratio was within the interval (0.5, 2); GMR = 1.07, 95% CI 2-sided [0.88 to 1.31] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Clostridium Difficile Vaccine: Lot 2 vs Clostridium Difficile Vaccine: Lot 3; Toxin B; Test type: Equivalence — Equivalence was established if the 95% confidence interval of GMC ratio was within the interval (0.5, 2); GMR = 1.01, 95% CI 2-sided [0.83 to 1.23] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 1
Description: Local reactions included pain at injection site, redness and swelling. These were recorded by participants in an electronic diary (e-diary). Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity, grade 4: emergency room visit or hospitalization. Redness and swelling were measured and recorded in measuring device units. One measuring device unit= 0.5 centimeter (cm) and graded as mild: 2.5 to 5.0 cm, moderate: greater than (>) 5.0 to 10.0 cm, severe: >10.0 cm, Grade 4 indicated necrosis or exfoliative dermatitis for redness and necrosis for swelling. The maximum severity was defined as highest grading of each local reaction within 7 days of vaccination. Events were classified as Grade 4 based on study investigator's judgement.
Time Frame: Within 7 days after Vaccination 1 at Month 0
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Number analyzed (Participants) | 325 | 320 | 322 | 325
Percentage of participants
  Pain at injection site: Mild | 14.2 [10.6 to 18.4] | 15.9 [12.1 to 20.4] | 17.4 [13.4 to 22.0] | 4.9 [2.8 to 7.9]
  Pain at injection site: Moderate | 2.5 [1.1 to 4.8] | 0.3 [0.0 to 1.7] | 0.9 [0.2 to 2.7] | 0 [0.0 to 1.1]
  Pain at injection site: Severe | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Pain at injection site: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Redness: Mild | 0.6 [0.1 to 2.2] | 1.6 [0.5 to 3.6] | 2.2 [0.9 to 4.4] | 0.6 [0.1 to 2.2]
  Redness: Moderate | 0.6 [0.1 to 2.2] | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Redness: Severe | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Redness: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Swelling: Mild | 1.5 [0.5 to 3.6] | 0.9 [0.2 to 2.7] | 1.6 [0.5 to 3.6] | 0 [0.0 to 1.1]
  Swelling: Moderate | 0.9 [0.2 to 2.7] | 0.6 [0.1 to 2.2] | 0.3 [0.0 to 1.7] | 0.6 [0.1 to 2.2]
  Swelling: Severe | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0.6 [0.1 to 2.2] | 0 [0.0 to 1.1]
  Swelling: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]

3. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 2
Description: Local reactions included pain at injection site, redness and swelling. These were recorded by participants in an e-diary. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity, grade 4: emergency room visit or hospitalization. Redness and swelling were measured and recorded in measuring device units. One measuring device unit= 0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm, severe: >10.0 cm, Grade 4 indicated necrosis or exfoliative dermatitis for redness and necrosis for swelling. The maximum severity was defined as highest grading of each local reaction within 7 days of vaccination. Events were classified as Grade 4 based on study investigator's judgement.
Time Frame: Within 7 days after Vaccination 2 at Month 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Number analyzed (Participants) | 316 | 309 | 314 | 313
Percentage of participants
  Pain at injection site: Mild | 22.2 [17.7 to 27.1] | 26.9 [22.0 to 32.2] | 22.0 [17.5 to 27.0] | 4.2 [2.2 to 7.0]
  Pain at injection site: Moderate | 2.2 [0.9 to 4.5] | 2.9 [1.3 to 5.5] | 1.6 [0.5 to 3.7] | 0.3 [0.0 to 1.8]
  Pain at injection site: Severe | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Pain at injection site: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Redness: Mild | 3.5 [1.8 to 6.1] | 3.9 [2.0 to 6.7] | 1.3 [0.3 to 3.2] | 1.0 [0.2 to 2.8]
  Redness: Moderate | 1.9 [0.7 to 4.1] | 1.3 [0.4 to 3.3] | 1.3 [0.3 to 3.2] | 0.3 [0.0 to 1.8]
  Redness: Severe | 1.3 [0.3 to 3.2] | 0.6 [0.1 to 2.3] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Redness: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Swelling: Mild | 3.5 [1.8 to 6.1] | 3.9 [2.0 to 6.7] | 1.9 [0.7 to 4.1] | 0.3 [0.0 to 1.8]
  Swelling: Moderate | 2.5 [1.1 to 4.9] | 1.6 [0.5 to 3.7] | 1.6 [0.5 to 3.7] | 0 [0.0 to 1.2]
  Swelling: Severe | 0.9 [0.2 to 2.7] | 1.3 [0.4 to 3.3] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2]
  Swelling: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

4. Primary Outcome: Percentage of Participants Reporting Local Reactions by Maximum Severity Within 7 Days After Vaccination 3
Description: as for outcome 3
Time Frame: Within 7 days after Vaccination 3 at Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Number analyzed (Participants) | 293 | 295 | 298 | 303
Percentage of participants
  Pain at injection site: Mild | 22.5 [17.9 to 27.7] | 23.4 [18.7 to 28.6] | 27.9 [22.8 to 33.3] | 2.6 [1.1 to 5.1]
  Pain at injection site: Moderate | 1.7 [0.6 to 3.9] | 2.0 [0.7 to 4.4] | 1.3 [0.4 to 3.4] | 0.3 [0.0 to 1.8]
  Pain at injection site: Severe | 0 [0.0 to 1.3] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Pain at injection site: Grade 4 | 0 [0.0 to 1.3] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Redness: Mild | 2.4 [1.0 to 4.9] | 3.7 [1.9 to 6.6] | 2.0 [0.7 to 4.3] | 0.7 [0.1 to 2.4]
  Redness: Moderate | 1.0 [0.2 to 3.0] | 2.0 [0.7 to 4.4] | 0.7 [0.1 to 2.4] | 0.3 [0.0 to 1.8]
  Redness: Severe | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2]
  Redness: Grade 4 | 0 [0.0 to 1.3] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Swelling: Mild | 2.4 [1.0 to 4.9] | 5.8 [3.4 to 9.1] | 3.7 [1.9 to 6.5] | 0.7 [0.1 to 2.4]
  Swelling: Moderate | 1.0 [0.2 to 3.0] | 2.7 [1.2 to 5.3] | 1.7 [0.5 to 3.9] | 0 [0.0 to 1.2]
  Swelling: Severe | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.9] | 0.3 [0.0 to 1.8]
  Swelling: Grade 4 | 0 [0.0 to 1.3] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

5. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 1
Description: Systemic events included fever, fatigue, headache, joint pain, muscle pain and vomiting. These were recorded by participants in an e-diary. Fever was categorized as: mild: (38.0 to 38.4 degree Celsius [deg C]), moderate: (38.5 to 38.9 deg C), severe (39.0 to 40.0 deg C), grade 4: >40 deg C. Fatigue, headache, joint pain and muscle pain were graded as mild: did not interfere with activity, moderate: some interference with activity, severe: prevented daily activity, grade 4: emergency room visit or hospitalization. Vomiting was graded as mild: 1 to 2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration, grade 4: emergency room visit or hospitalization for hypotensive shock. The maximum severity was defined as highest grading of each systemic event within 7 days of vaccination. Events were classified as Grade 4 based on study investigator's judgement.
Time Frame: Within 7 days after Vaccination 1 at Month 0
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Number analyzed (Participants) | 325 | 320 | 322 | 325
Percentage of participants
  Fever: 38.0-38.4 deg C | 0.9 [0.2 to 2.6] | 0.6 [0.1 to 2.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Fever: 38.5-38.9 deg C | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Fever: 39.0-40.0 deg C | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Fever: >40 deg C | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Fatigue: Mild | 11.7 [8.3 to 15.5] | 10.9 [7.6 to 14.7] | 14.0 [10.2 to 17.9] | 8.3 [5.4 to 11.6]
  Fatigue: Moderate | 12.0 [8.5 to 15.8] | 9.1 [6.1 to 12.6] | 9.6 [6.5 to 13.1] | 10.2 [7.0 to 13.7]
  Fatigue: Severe | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1] | 0.9 [0.2 to 2.6] | 0 [0.0 to 1.1]
  Fatigue: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Headache: Mild | 13.2 [9.6 to 17.1] | 11.3 [7.9 to 15.0] | 6.5 [4.0 to 9.6] | 7.7 [4.9 to 10.9]
  Headache: Moderate | 3.7 [1.9 to 6.3] | 4.1 [2.1 to 6.7] | 5.3 [3.0 to 8.2] | 3.4 [1.7 to 5.9]
  Headache: Severe | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0.6 [0.1 to 2.2] | 0.3 [0.0 to 1.7]
  Headache: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Joint pain: Mild | 4.9 [2.8 to 7.8] | 3.8 [1.9 to 6.4] | 4.0 [2.1 to 6.7] | 2.2 [0.9 to 4.3]
  Joint pain: Moderate | 3.7 [1.9 to 6.3] | 2.8 [1.3 to 5.2] | 4.3 [2.4 to 7.1] | 3.1 [1.5 to 5.5]
  Joint pain: Severe | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Joint pain: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Muscle pain: Mild | 4.6 [2.6 to 7.4] | 3.1 [1.5 to 5.6] | 3.4 [1.7 to 5.9] | 5.2 [3.0 to 8.1]
  Muscle pain: Moderate | 4.6 [2.6 to 7.4] | 4.7 [2.6 to 7.5] | 3.1 [1.5 to 5.5] | 4.6 [2.6 to 7.4]
  Muscle pain: Severe | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Muscle pain: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Vomiting: Mild | 0.3 [0.0 to 1.7] | 0.9 [0.2 to 2.7] | 0.9 [0.2 to 2.6] | 0.3 [0.0 to 1.7]
  Vomiting: Moderate | 0.9 [0.2 to 2.6] | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7]
  Vomiting: Severe | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Vomiting: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 2
Description: Systemic events included fever, fatigue, headache, joint pain, muscle pain and vomiting. These were recorded by participants in an e-diary. Fever was categorized as: mild: (38.0 to 38.4 deg C), moderate: (38.5 to 38.9 deg C), severe (39.0 to 40.0 deg C), grade 4: >40 deg C. Fatigue, headache, joint pain and muscle pain were graded as mild: did not interfere with activity, moderate: some interference with activity, severe: prevented daily activity, grade 4: emergency room visit or hospitalization. Vomiting was graded as mild: 1 to 2 times in 24 hours, moderate: >2 times in 24 hours, severe: required intravenous hydration, grade 4: emergency room visit or hospitalization for hypotensive shock. The maximum severity was defined as highest grading of each systemic event within 7 days of vaccination. Events were classified as Grade 4 based on study investigator's judgement.
Time Frame: Within 7 days after Vaccination 2 at Month 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Number analyzed (Participants) | 316 | 309 | 314 | 313
Percentage of participants
  Fever: 38.0-38.4 deg C | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Fever: 38.5-38.9 deg C | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Fever: 39.0-40.0 deg C | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Fever: >40 deg C | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Fatigue: Mild | 10.4 [7.2 to 14.1] | 11.0 [7.5 to 14.7] | 10.8 [7.5 to 14.6] | 4.8 [2.6 to 7.6]
  Fatigue: Moderate | 9.5 [6.4 to 13.0] | 8.7 [5.7 to 12.2] | 10.2 [7.0 to 13.9] | 6.4 [3.8 to 9.4]
  Fatigue: Severe | 1.3 [0.3 to 3.1] | 0.6 [0.1 to 2.3] | 0.6 [0.1 to 2.2] | 1.0 [0.2 to 2.7]
  Fatigue: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Headache: Mild | 8.2 [5.3 to 11.6] | 10.4 [7.0 to 14.0] | 8.6 [5.7 to 12.1] | 5.8 [3.3 to 8.7]
  Headache: Moderate | 4.4 [2.4 to 7.2] | 2.3 [0.9 to 4.5] | 4.8 [2.7 to 7.6] | 3.2 [1.5 to 5.6]
  Headache: Severe | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7] | 0.6 [0.1 to 2.2] | 0 [0.0 to 1.1]
  Headache: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Joint pain: Mild | 4.7 [2.6 to 7.6] | 5.2 [2.9 to 8.1] | 3.2 [1.5 to 5.7] | 1.6 [0.5 to 3.6]
  Joint pain: Moderate | 4.4 [2.4 to 7.2] | 3.9 [2.0 to 6.5] | 2.9 [1.3 to 5.3] | 2.2 [0.9 to 4.4]
  Joint pain: Severe | 0.6 [0.1 to 2.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Joint pain: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Muscle pain: Mild | 3.8 [1.9 to 6.4] | 4.5 [2.4 to 7.3] | 3.8 [2.0 to 6.5] | 2.2 [0.9 to 4.4]
  Muscle pain: Moderate | 5.4 [3.1 to 8.3] | 3.2 [1.5 to 5.7] | 4.5 [2.4 to 7.3] | 1.3 [0.3 to 3.1]
  Muscle pain: Severe | 0.6 [0.1 to 2.2] | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Muscle pain: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Vomiting: Mild | 0.9 [0.2 to 2.7] | 0 [0.0 to 1.2] | 1.3 [0.3 to 3.2] | 0.6 [0.1 to 2.2]
  Vomiting: Moderate | 0 [0.0 to 1.1] | 0.3 [0.0 to 1.7] | 0.3 [0.0 to 1.7] | 0 [0.0 to 1.1]
  Vomiting: Severe | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]
  Vomiting: Grade 4 | 0 [0.0 to 1.1] | 0 [0.0 to 1.2] | 0 [0.0 to 1.1] | 0 [0.0 to 1.1]

7. Primary Outcome: Percentage of Participants Reporting Systemic Events by Maximum Severity Within 7 Days After Vaccination 3
Description: as for outcome 6
Time Frame: Within 7 days after Vaccination 3 at Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine: Lot 1 | Clostridium Difficile Vaccine: Lot 2 | Clostridium Difficile Vaccine: Lot 3 | Placebo
Number analyzed (Participants) | 293 | 295 | 298 | 303
Percentage of participants
  Fever: 38.0-38.4 deg C | 0.3 [0.0 to 1.8] | 0.3 [0.0 to 1.8] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2]
  Fever: 38.5-38.9 deg C | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0.7 [0.1 to 2.3]
  Fever: 39.0-40.0 deg C | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Fever: >40 deg C | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Fatigue: Mild | 10.6 [7.0 to 14.1] | 8.5 [5.4 to 11.9] | 10.4 [7.0 to 14.0] | 5.0 [2.8 to 7.9]
  Fatigue: Moderate | 10.6 [7.0 to 14.1] | 7.8 [4.8 to 11.1] | 5.7 [3.3 to 8.7] | 8.6 [5.6 to 12.1]
  Fatigue: Severe | 0 [0.0 to 1.2] | 1.0 [0.2 to 2.8] | 1.0 [0.2 to 2.8] | 0 [0.0 to 1.2]
  Fatigue: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Headache: Mild | 12.6 [8.7 to 16.3] | 8.8 [5.6 to 12.2] | 7.0 [4.3 to 10.3] | 5.9 [3.5 to 9.1]
  Headache: Moderate | 3.4 [1.6 to 5.9] | 3.7 [1.8 to 6.4] | 2.7 [1.1 to 5.1] | 1.7 [0.5 to 3.7]
  Headache: Severe | 0.7 [0.1 to 2.3] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Headache: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Joint pain: Mild | 2.0 [0.7 to 4.2] | 2.7 [1.1 to 5.1] | 2.7 [1.1 to 5.1] | 3.0 [1.3 to 5.5]
  Joint pain: Moderate | 2.7 [1.1 to 5.1] | 1.7 [0.5 to 3.8] | 2.7 [1.1 to 5.1] | 0.7 [0.1 to 2.3]
  Joint pain: Severe | 0.3 [0.0 to 1.8] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Joint pain: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Muscle pain: Mild | 3.1 [1.4 to 5.5] | 3.1 [1.4 to 5.5] | 5.0 [2.8 to 7.9] | 2.6 [1.1 to 5.1]
  Muscle pain: Moderate | 2.4 [0.9 to 4.7] | 2.0 [0.7 to 4.2] | 3.0 [1.3 to 5.5] | 1.7 [0.5 to 3.7]
  Muscle pain: Severe | 0.3 [0.0 to 1.8] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Muscle pain: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Mild | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0.7 [0.1 to 2.3]
  Vomiting: Moderate | 0.7 [0.1 to 2.3] | 0.7 [0.1 to 2.3] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Severe | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Grade 4 | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

8. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Through 1 Month After Last Study Vaccination
Description: An AE was defined as any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and all non-serious adverse events (NSAEs). Only AEs and NSAEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Day 1 to 1 month after last vaccination (Up to Month 7)
Population: Safety analysis population included all participants who received at least 1 dose of the investigational product. Pooled data for Clostridium difficile vaccine (lot 1+lot 2+lot 3) is reported for this outcome measure as pre-specified in the statistical analysis plan.
Measure: Number; unit: Percentage of participants
Groups:
- Clostridium Difficile Vaccine (Pooled Lots): Participants received Clostridium difficile vaccine (200 microgram total toxoid per dose) Lot 1, Lot 2 or Lot 3 intramuscularly at Months 0, 1 and 6.
Arm/Group | Clostridium Difficile Vaccine (Pooled Lots) | Placebo
Number analyzed (Participants) | 983 | 331
Percentage of participants
  Any AEs | 35.5 | 33.5
  NSAEs | 34.1 | 31.7

9. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: From Day 1 to 1 month after last vaccination (Up to Month 7)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Clostridium Difficile Vaccine (Pooled Lots) | Placebo
Number analyzed (Participants) | 983 | 331
Percentage of participants | 4.2 | 4.5

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events (systematic assessment): within 7 days after vaccination. SAEs and other AEs: From Day 1 to 1 month after last vaccination (Up to Month 7)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis population was evaluated. Pooled data for Clostridium difficile vaccine (lot 1+lot 2+lot 3) is reported as pre-specified in the statistical analysis plan.
Arm/Group | Clostridium Difficile Vaccine (Pooled Lots) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/983 | 2/331
Serious Adverse Events (participants affected / at risk) | 41/983 | 15/331
Other Adverse Events (participants affected / at risk) | 694/983 | 175/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clostridium Difficile Vaccine (Pooled Lots) (N=983) | Placebo (N=331)
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Foot operation (Surgical and medical procedures) | 0 | 1
Hypertensive emergency (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clostridium Difficile Vaccine (Pooled Lots) (N=983) | Placebo (N=331)
Diarrhoea (Gastrointestinal disorders) | 11 | 3
Vomiting (VOMITING) (Gastrointestinal disorders) | 25 | 6
Fatigue (FATIGUE) (General disorders) | 369 | 96
Fatigue (General disorders) | 5 | 4
Injection site erythema (REDNESS) (General disorders) | 93 | 7
Injection site pain (PAIN) (General disorders) | 413 | 34
Injection site swelling (SWELLING) (General disorders) | 103 | 5
Pyrexia (FEVER) (General disorders) | 12 | 2
Bronchitis (Infections and infestations) | 16 | 3
Cellulitis (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 4 | 5
Nasopharyngitis (Infections and infestations) | 13 | 5
Sinusitis (Infections and infestations) | 11 | 2
Upper respiratory tract infection (Infections and infestations) | 40 | 13
Fall (Injury, poisoning and procedural complications) | 8 | 4
Procedural pain (Injury, poisoning and procedural complications) | 12 | 2
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 162 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 183 | 49
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4
Headache (HEADACHE) (Nervous system disorders) | 276 | 64
Hypertension (Vascular disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03579459/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03579459/SAP_001.pdf